CLINICAL TRIAL: NCT01717274
Title: Hot Saline Irrigation vs Room Temperature Saline Irrigation in the Control of Intraoperative Bleeding During Functional Endoscopic Sinus Surgery (FESS)
Brief Title: Hot Saline Irrigation Study
Acronym: HSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Paul's Hospital, Canada (Other)
Responsible Party: Principal Investigator, Amin Javer, Principal Investigator, St. Paul's Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: HSI-2012
Record Dates: First submitted 2012-10-26; First posted 2012-10-30 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Sinusitis
Keywords: Functional Endoscopic Sinus Surgery; Hot water irrigation
MeSH Terms: conditions — Sinusitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hot saline irrigation (Experimental): Hot saline is prepared by first placing 2 litres of sterile normal saline (0.9%) into a basin (IntraTemp Therma BasinTM) that is wrapped in a sterile disposable drape (IntraTemp Therma Basin DrapeTM). The basin is then placed in a medical grade warmer (IntraTemp Fluid Warming SystemTM). The warmer is set to heat the saline up to a temperature of 50 degrees Celsius. An external digital thermometer is placed in the saline at all times to ensure that the temperature is between 45-50 degrees.
  Interventions: Procedure: Hot saline irrigation
- Room temperature saline irrigation (No Intervention): Room temperature saline is prepared in the same manner as the experimental arm except that the warmer is switched off and the temperature of the saline in the basin is left to equilibrate to the temperature of the operating room.

INTERVENTIONS:
Procedure: Hot saline irrigation — The surgical field is flushed with 20 cc of hot saline (45-50 degrees Celsius) at five minutes intervals. This is in contrast to the standard of care, room temperature (20-25 degrees Celsius) saline irrigation.
  Other Names: HSI
  Arms: Hot saline irrigation

SUMMARY:
Many methods have been used to reduce bleeding during sinus surgery (FESS) in order to allow for the best surgical view and to reduce risk while in surgery.

Warm irrigation fluid is believed to accelerate the clotting mechanism in the human body. The investigators would like to determine if hot saline irrigation (HSI) compared to room temperature saline irrigation (RTSI) can control bleeding during FESS.

The hypothesis is that HSI is more effective than RTSI in reducing intraoperative bleeding during FESS.

DETAILED DESCRIPTION:
Background and Significance:

Functional endoscopic sinus surgery (FESS) is a minimally invasive surgery to relieve obstruction and to facilitate drainage and ventilation of the paranasal sinuses. It is a common rhinologic procedure that is safe, comfortable and allows quick patient recovery. As the paranasal sinuses have complex anatomy and are surrounded by important structures, there are risks of serious orbital and intracranial injuries. These risks are increased if visualization during surgery is impaired with bleeding. The endoscopically magnified operative field in sinus surgery makes even a small amount of bleeding a potentially significant hindrance. Hence, numerous methods to reduce intraoperative bleeding during FESS have been described. These include the use of preoperative nasal decongestion (such as topical oxymetazoline, cocaine and adrenaline), preoperative oral tranexamic acid, intraoperative injection of the lateral nasal wall with lidocaine and adrenaline and intraoperative controlled hypotension (using total intravenous anaesthesia and B-blockers) as well as the head up position during surgery. The success rates of these methods have been variable and some of these techniques are associated with adverse cardiopulmonary events.1-7 Visual compromise secondary to bleeding remains a problem during FESS and the ideal method to reduce intraoperative bleeding remains elusive.

Hot water irrigation (HWI) was first used by obstetricians in controlling postpartum bleeding over a hundred years ago.8 Its use in the control of intractable epistaxis was first described by Guice in 1878.9 In a histological study of nasal mucosa of rabbits irrigated with hot water, Stangerup and Thomsen found that temperatures of up to 50 degrees Celsius produces vasodilation and edema of the nasal mucosa without necrosis. They postulated that mucosal edema leads to compression of the bleeding vessels and may trigger and accelerate the clotting cascade.10 Stangerup et al found that in their series of 122 patients, posterior epistaxis was controlled in 55% of patients treated with HWI compared to 44% in the group treated with nasal packing.11 Novoa and Schlegel-Wagner subsequently showed that 82% of patients with intractable posterior epistaxis can be arrested with HWI.12 HWI has also led to reduced hospital stay, reduced number of surgical procedures, less pain and less nasal trauma. As continuous exposure of the nasal mucosa to pure water for 30 minutes has been shown by an in-vitro study to cause severe damage to the epithelial cells, we have decided to use hot normal saline in our study.13 Although hot saline irrigation (HSI) has been used in FESS and endoscopic skull base surgery, there are currently no reports in the English literature on its effectiveness.

Aim:

To assess the effectiveness of hot saline irrigation (HSI) compared to room temperature saline irrigation (RTSI) in the control of intraoperative bleeding during FESS.

Hypothesis:

HSI is more effective than RTSI in reducing intraoperative bleeding during FESS

Experimental design and methods:

Target population:

Patients are recruited from the St. Paul's Sinus Centre at St. Paul's hospital in Vancouver, Canada.

Sample size: 60 patients (30 patients in each arm)

Preoperative data collection:

The following data is collected preoperatively:

1. Patient's demographics (age, sex, race)
2. Preoperative Lund and Mackay Score
3. Presence of polyps

Research design:

Double blind randomized control trial

Preoperative:

All patients are treated with a one-week course of prednisone 20mg once a day and oral antibiotics (clavulin or clindamycin if penicillin) prior to surgical intervention.

Intraoperative:

Procedure:

Using a closed envelope system, patients enrolled in the study are randomized to receive either HSI (defined as temperatures of 45-50 degrees Celsius) or RTSI (defined as temperature of the operating room). Both the patient and the surgeon are blinded to the temperature of the irrigation fluid used during surgery. After randomization, a nominated research assistant will receive instructions to prepare the hot or room temperature saline solution.

Experimental arm:

Hot saline is prepared by first placing 2 litres of sterile normal saline (0.9%) into a basin (IntraTemp Therma BasinTM) that is wrapped in a sterile disposable drape (IntraTemp Therma Basin DrapeTM). The basin is then placed in a medical grade warmer (IntraTemp Fluid Warming SystemTM). The warmer is set to heat the saline up to a temperature of 50 degrees Celsius. An external digital thermometer is placed in the saline at all times to ensure that the temperature is between 45-50 degrees.

Control arm:

Room temperature saline is prepared in the same manner except that the warmer is switched off and the temperature of the saline in the basin is left to equilibrate to the temperature of the operating room.

In both arms, a 60 cc syringe attached to an olive tip long curve suction is used to draw the irrigation fluid from the basin. The surgical field is flushed with 20 cc of hot or room temperature saline at five minutes intervals by a research assistant. Additional flushes with hot or room temperature saline can be administered in between the five-minute intervals upon request by the surgeon. The degree of bleeding in the surgical field is scored by the operating surgeon using the validated Boezaart and van der Merwe Grading System14. This 0 to 5-point scale will be used to outline the amount of suction required to rid the area of blood disrupting vision. A score of 0 is given for an area with no bleeding, 1 for slight bleeding with no suction required, 2 for slight bleeding requiring suction, 3 for moderate bleeding which improves for several seconds once suction has occurred, 4 for moderate bleeding which restarts directly after suctioning and 5 for severe bleeding which occurs faster then can be removed14. Surgical field of view will be assessed and scored every 15 minutes for the duration of the surgery. At the end of the procedure, the estimated blood loss is calculated by subtracting the total amount of irrigation fluid used from the fluid in the suction bottle. The total amount of HSI or RTSI administered and time of surgery are documented.

Surgery:

Patients are placed under general anesthesia and intubated with endotracheal tubes. Immediately after general anesthesia, both nasal cavities are packed with neuropatties soaked with Otrivin (xylometazolin 0.05%). The patients' heads are elevated 15 degrees up. The image guided system is set up and each nasal cavity is examined with a 0 degree endoscope. A 10 cm merocel is cut into a third of its normal size and inserted to the back of the nasopharynx, to prevent blood from flowing into the oropharynx and larynx. An artery forceps is clipped onto the merocel string to prevent dislodgement of the merocel into the larynx or oropharynx. FESS is performed using the technique described by Messerklinger15 and with a microdebrider when deemed necessary. The extent of the operation depends on the severity of the disease seen on the pre-operative CT scan of the paranasal sinus.

Data collection and analysis:

This is a pilot study; hence the statistical analysis will be completed at the end of the study.

Clinically significant change in intra-operative bleeding will be defined as a change in Boezaart scoring by 20%, or one point in relation to the scale. All data collected for this study will be gathered in a password protected Microsoft Excel spreadsheet file. Each patient will be assigned unique identification allowing for no patient data to be recorded. The Microsoft Excel database will include:

* Age
* Sex
* Pre-existing health conditions
* Current medications
* Lund-Kennedy CT score
* CRS with or without polyposis
* Primary or revision surgery
* Anesthesia infusion
* MAP (15 minute intervals)
* Pulse rate (15 minute intervals)
* Endoscopic surgical field scores (15 minute intervals)
* Intra-operative complications
* Microdebrider usage
* Total blood loss
* Total time of surgery
* Total saline irrigation used

Risk:

The use of nasal irrigation of up to 50 degrees Celsius have been shown to be safe on the epithelium of rabbit nasal mucosa studied in-vitro.10 In addition, studies have shown that irrigation of the human nasal mucosa with temperatures of up to 50 degrees Celsius did not result in any complications.11,12 Hot saline irrigation has been widely used for skull base and endoscopic sinus surgery for many years with no known reported complication in the English literature.

Difficulties and limitation:

Patient recruitment:

Based on the surgical volume at St Paul's Sinus Centre, we do not foresee any difficulties in achieving the target sample size. The St Paul's Sinus Centre is actively involved in research. Many of our patients are aware of this and are keen to participate in and contribute to medical research.

Achieving the desired temperature:

The exact temperature of 50 degrees Celsius is difficult to achieve. Hence we defined our HSI with a range of temperature of 45-50 degrees Celsius

ELIGIBILITY:
Inclusion Criteria:

* Patients with American Society of Anesthesiologist (ASA) classification <2
* Patients with chronic or recurrent sinusitis (as defined by the American Academy of Otolaryngology) with or without nasal polyposis refractory to medical treatment

Exclusion Criteria:

* Patients with a history of coagulation disorders
* Patients with severe ischemic heart disease (IHD), pulmonary and renal disease
* Patients with tumours or vascular anomalies
* Patients with cystic fibrosis, allergic fungal sinusitis and Wegener's granulomatosis
* Patients who are unable to speak, read and write English

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-11; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
The Boezaart and van der Merwe intraoperative surgical field scale | Every 15 minutes for the duration of surgery..
  The Boezaart intra-operative surgical field scale will be used to grade the level of bleeding during surgery. This 0 to 5-point scale will be used to outline the amount of suction required to rid the area of blood disrupting vision. A score of 0 is given for an area with no bleeding, 1 for slight bleeding with no suction required, 2 for slight bleeding requiring suction, 3 for moderate bleeding which improves for several seconds once suction has occurred, 4 for moderate bleeding which restarts directly after suctioning and 5 for severe bleeding which occurs faster then can be removed

SECONDARY OUTCOMES:
Total Estimated Blood Loss | Duration of surgery
  Total blood loss will be recorded over the duration of surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Amin R Javer, MD, FRCSC, FARS, Principal Investigator — St Pauls Hospital
Locations (1):
- E.N.T. Clinic, St. Paul's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Riegle EV, Gunter JB, Lusk RP, Muntz HR, Weiss KL. Comparison of vasoconstrictors for functional endoscopic sinus surgery in children. Laryngoscope. 1992 Jul;102(7):820-3. doi: 10.1288/00005537-199207000-00012. PMID 1614253
- [Background] Yaniv E, Shvero J, Hadar T. Hemostatic effect of tranexamic acid in elective nasal surgery. Am J Rhinol. 2006 Mar-Apr;20(2):227-9. PMID 16686395
- [Background] Tirelli G, Bigarini S, Russolo M, Lucangelo U, Gullo A. Total intravenous anaesthesia in endoscopic sinus-nasal surgery. Acta Otorhinolaryngol Ital. 2004 Jun;24(3):137-44. PMID 15584584
- [Background] Higgins TS, Hwang PH, Kingdom TT, Orlandi RR, Stammberger H, Han JK. Systematic review of topical vasoconstrictors in endoscopic sinus surgery. Laryngoscope. 2011 Feb;121(2):422-32. doi: 10.1002/lary.21286. Epub 2011 Jan 13. PMID 21271600
- [Background] Stangerup SE, Dommerby H, Siim C, Kemp L, Stage J. New modification of hot-water irrigation in the treatment of posterior epistaxis. Arch Otolaryngol Head Neck Surg. 1999 Jun;125(6):686-90. doi: 10.1001/archotol.125.6.686. PMID 10367928
- [Background] Novoa E, Schlegel-Wagner C. Hot water irrigation as treatment for intractable posterior epistaxis in an out-patient setting. J Laryngol Otol. 2012 Jan;126(1):58-60. doi: 10.1017/S002221511100243X. Epub 2011 Sep 5. PMID 21888749
- [Background] Javer AR, Gheriani H, Mechor B, Flamer D, Genoway K, Yunker WK. Effect of intraoperative injection of 0.25% bupivacaine with 1:200,000 epinephrine on intraoperative blood loss in FESS. Am J Rhinol Allergy. 2009 Jul-Aug;23(4):437-41. doi: 10.2500/ajra.2009.23.3339. PMID 19671263
- [Derived] Gan EC, Alsaleh S, Manji J, Habib AR, Amanian A, Javer AR. Hemostatic effect of hot saline irrigation during functional endoscopic sinus surgery: a randomized controlled trial. Int Forum Allergy Rhinol. 2014 Nov;4(11):877-84. doi: 10.1002/alr.21376. Epub 2014 Aug 18. PMID 25137523